CLINICAL TRIAL: NCT01490385
Title: The Effect of Light Emitting Diode Phototherapy on the Rate of Orthodontic Tooth Movement - A Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bryan Tompson (Other)
Responsible Party: Sponsor-Investigator, Bryan Tompson, Head, Discipline of Orthodontics, University of Toronto
Organization: University of Toronto (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 11-12-2
Record Dates: First submitted 2011-11-10; First posted 2011-12-13 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: The Rate or Orthodontic Tooth Movement

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LED Phototherapy (Active Comparator): LED phototherapy will be delivered transdermally via an extra-oral device and in a split mouth manner (half of the dental arch).
  Interventions: Device: LED Phototherapy
- Control: conventional orthodontic tooth movement (No Intervention)

INTERVENTIONS:
Device: LED Phototherapy
  Other Names: Device manufactured by Biolux Research Ltd
  Arms: LED Phototherapy

SUMMARY:
LED Phototherapy will increase the velocity of Orthodontic tooth movement.

ELIGIBILITY:
Inclusion Criteria:

* bilaterally symmetric extraction of premolar teeth with residual extraction spaces large enough to ensure space closure is not complete prior to the subsequent orthodontic appointment
* no medicines or systemic illness
* full banding/bonding of teeth

Exclusion Criteria:

* pregnant
* non-extraction treatment
* systemic illness
* prior orthodontic treatment

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Extraction space size | T0, T1, T2
  T0=the start of active extraction space closure T1=3-7 weeks after T0 T2=4-7 weeks after T1

CONTACTS AND LOCATIONS:
Overall Officials: Bryan D Tompson, DDS, DipPaedo, DipOrtho, FRCDC, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Faculty of Dentistry, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Chung SE, Tompson B, Gong SG. The effect of light emitting diode phototherapy on rate of orthodontic tooth movement: a split mouth, controlled clinical trial. J Orthod. 2015;42(4):274-83. doi: 10.1179/1465313315Y.0000000013. Epub 2015 Jul 28. PMID 26216550